CLINICAL TRIAL: NCT05695274
Title: Effect of Progressive Muscle Relaxation Exercises on Pain, Kinesiophobia and Functional Status in Fibromyalgia Patients
Brief Title: Progressive Muscle Relaxation Exercises on Pain, Kinesiophobia and Functional Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cemile KÜTMEÇ YILMAZ, Principal Investigator, Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2022/14-05
Record Dates: First submitted 2023-01-05; First posted 2023-01-25 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): To examine the effects of progressive muscle relaxation exercises on pain, kinesiophobia and functional status in fibromyalgia patients.
  Interventions: Behavioral: Progressive muscle relaxation exercise
- Control group (No Intervention): Control group; routine care and treatment will be applied.

INTERVENTIONS:
Behavioral: Progressive muscle relaxation exercise — Experimental group Fibromyalgia patients will be provided with progressive relaxation exercises twice a week. Progressive relaxation technique includes stretching and relaxing the bigmuscle groups (hands, arms, neck, shoulders, face, chest, abdomen,hip, feet andfingers) in the human body on purpose. When steps ofProgressive Relaxation Exercises are analyzed, it is observed thatlearning how to take correct and deep breaths is the most impor-tant step towards learning relaxation.
  Arms: Experimental group

SUMMARY:
Relaxation techniques are a non-pharmacological therapy option applied to alleviate the symptoms of many different chronic diseases. It has been reported in the literature that PMR is effective on pain, fatigue and stress symptoms in fibromyalgia patients. No study has been found examining the effect of PMR on kinesiophobia and functional status in FM. This study was planned to examine the effect of progressive muscle relaxation exercises on pain, kinesiophobia and functional status in fibromyalgia patients.

DETAILED DESCRIPTION:
Fibromyalgia (FM), which is a chronic pain disorder, is a difficult disease to treat, and it is stated that a multidisciplinary approach is required in its treatment rather than a single treatment method. Approaches that consider optimal symptom management and functional status in treatment, include non-pharmacological methods in addition to pharmacological treatment, and include psychosocial and behavioral methods are recommended. Non-pharmacological methods that have proven their effectiveness in FM treatment include aerobic exercise, patient education, cognitive therapies, balneotherapy, and physical therapy agents. One of the methods that can be applied in patients with FM is progressive muscle relaxation (PMR) exercises. PMR is an easy, low-cost, and side-effect-free relaxation technique. PMR helps individuals feel calmer and more relaxed through sequential muscle tension and relaxation. It has been reported in the literature that PMR is effective on pain, fatigue and stress symptoms in fibromyalgia patients. No study has been found examining the effect of PMR on kinesiophobia and functional status in FM. Therefore, this study was planned to examine the effect of progressive muscle relaxation exercises on pain, kinesiophobia and functional status in fibromyalgia patients.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 years of age
* Having been diagnosed with fibromiyalgia for at least 6 months ago.
* Having no mental disability

Exclusion Criteria:

* Individuals receiving another complementary and integrative treatment
* Individuals who have done progressive muscle relaxation exercise before.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Progressive muscle relaxation exercise changes pain | The pain scores of the patients will be measured before the PMR application and at the end of the PMR application (at the end of the 8th week) two days a week for the 8th week using the visual pain scale. The pain score is min 1 - max 10.
  Visual Pain Scale
Progressive muscle relaxation exercise changes kinesiophobia | The Kinesiophobia scores of patients will be measured before the PMR application and at the end of the PMR application (at the end of the 8th week) two days a week for the 8th week. A total of 17-68 points are obtained from the scale.
  Tampa Scale for Kinesiophobia
Progressive muscle relaxation exercise changes functional status | The functional status scores of patients will be measured before the PMR application and at the end of the PMR application (at the end of the 8th week) two days a week for the 8th week. A high score indicates increased disability due to FM.
  Revised Fibromyalgia Impact Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: CEMİLE KÜTMEÇ YILMAZ, Principal Investigator — Aksaray University, Faculty of Health Science, Nursing Department, Turkey
Locations (2):
- Turkey (Türkiye) (2):
  - Cemile KÜTMEÇ YILMAZ, Merkez, Aksaray
  - Aksaray University Health Science Faculty, Aksaray

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakoyun A, Kutmec Yilmaz C, Sayin Kasar K. Are Progressive Muscle Relaxation Exercises Effective on Pain, Kinesiophobia, and Functional Status in Fibromyalgia Patients? A Randomized Controlled Trial. Res Nurs Health. 2026 Feb;49(1):9-18. doi: 10.1002/nur.70029. Epub 2025 Nov 14. PMID 41235733